CLINICAL TRIAL: NCT02150252
Title: Randomized, Double Blind, Placebo Control Trial to Evaluate the Efficacy of Bu-Yang-Huan-Wu Tang（BYHWT）on Ischemic Stroke
Brief Title: Evaluate the Efficacy of Bu-Yang- Huan-Wu Tang（BYHWT）on Ischemic Stroke
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH102-REC1-122
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Ischemic Stroke
Keywords: Clinical trial; Ischemic stroke; Bu-Yang-Huan-Wu Tang (BYHWT）; Gait parameter; Quality of life
MeSH Terms: conditions — Ischemic Stroke | interventions — bu-yang-huan-wu-tang

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- BY HWT，placebo-BY HWT ， Gait parameter (Experimental)
  Interventions: Drug: Bu-Yang-Huan-Wu Tang

INTERVENTIONS:
Drug: Bu-Yang-Huan-Wu Tang — control group,Recruited patients should be received the placebo-BYHWT 3.0 g TID every day for continuously 6 weeks except ordinary medical care; 2) treatment group, the method is identical control group

SUMMARY:
* Clinical trial; Ischemic stroke; Bu-Yang-Huan-Wu Tang （BYHWT）; Gait parameter; Quality of life Stroke is the third of ten causing death disease constantly, and it also is third of consuming healthy insurance budget. There is 17,000 peoples disable due to stroke every year in Taiwan. Although ischemic stroke patient may use t-PA intravenously treatment within 3 hrs after stroke onset in modern medicine, and no others method may effect to treat ischemic stroke patients, thus, the study about stroke is an important issue. Bu-Yang- Huan-Wu Tang (BYHWT) has been became a main stream for the treatment of stroke after Qing dynasty Wang Qing-Ren theory that is BYHWT may treat stroke due to pattern of qi stagnation and blood stasis in traditional Chinese medicine. A number of researches report that BYHWT can reduce blood viscosity, anti-inflammation, enhancing neuronal regeneration and angiogenesis, but above-mentioned about BYHWT limit in the level of animal study and the scientific evidence is insufficiency in human trial. Therefore, the purpose of the present study was to investigate the therapeutic effect of BYHWT treating ischemic stroke by using a strict clinical trial.
* We designed a randomized, double blind, placebo-controlled study to assess the therapeutic effect of BYHWT treating ischemic stroke. The study expects to finish the assessment of 120 patients with ischemic stroke in three years. The study divided into: 1) control group, receive placebo-BYHWT 3.0 g TID every day for continuously 6 weeks except ordinary medical care; 2) treatment group, the method is identical control group, but receive BYHWY. The main outcome was according to the changes of gait parameter including Speed, Cadence, Strike length, Gait cycle and Double support; and secondary outcome including the changes of Functional independence measurement scores and Barthel index scores, Ten Meters Walk Test, Short Physical Performance Batter, Berg Balance Test and WHO quality of life-brief (Taiwan Brief).
* We predict the results of the present can provide scientific evidence to proof BYHWT can improve neurological deficit and also can improve quality of life in patients with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≧40 and ≦75
2. Stroke is first time
3. Between 15 and 90 day after stroke onset
4. NIHSS score between 5 and 20
5. NIHSS: 6th item, motor function (lower extremities) ≦3
6. Walking is at least 10 meters.

Exclusion Criteria:

1. Intake anticoagulant agent within one week, such as Heparin, warfarin etc.
2. NIHSS: 6th item, motor function (lower extremities) = 0 (lift 30 degree more than 5 second in supine position)
3. Cannot intake food from oral or intake food complete depend on helper
4. Acute stroke onset within 14 days
5. Gait disturbance due to other factor, such as Parkinson disease, spinal injury, knee joint disorders etc.
6. Cerebellar stroke
7. Pregnancy or lactation
8. Over irritability or anxiety results in cannot assessment
9. Severe traumatic injury or head surgery history
10. Stroke due to cerebral venous thrombosis
11. Systemic disease such as uremia, chronic obstructive pulmonary disorders, or heart failure NYHA ≧ (third degree: mild activity induces dyspnea; fourth degree: dyspnea feeling under rest state)
12. Severe psychiatric disorders such as depression, schizophrenia etc.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Gait parameter | 42days and 84days
  The main outcome was according to the changes of gait parameter including Speed, Cadence, Strike length, Gait cycle and Double support.

SECONDARY OUTCOMES:
Functional independence measurement scores and Barthel index scores, Ten Meters Walk Test, Short Physical Performance Batter, Berg Balance Test and WHO quality of life-brief (Taiwan Brief). | 42days and 84days

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan